CLINICAL TRIAL: NCT01355991
Title: Acute and Chronic Effects of an Anticholinergic Agent or a Long-Acting Beta 2 Agonist on Levels of Exhaled Nitric Oxide and Pulmonary Function in Persons With Tetraplegia
Brief Title: Effects of Anticholinergic or Long-Acting Beta 2 Agonist on FeNO and Pulmonary Function in SCI
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: James J. Peters Veterans Affairs Medical Center (U.S. Federal Agency)
Collaborators: Kessler Institute for Rehabilitation (Industry)
Responsible Party: Principal Investigator, Miroslav Radulovic, M.D., Staff Physician, James J. Peters Veterans Affairs Medical Center
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 01327
Record Dates: First submitted 2011-05-12; First posted 2011-05-19 (Estimated); Last update posted 2015-10-23 (Estimated); Status verified 2015-10

CONDITIONS: Spinal Cord Injury
Keywords: Spinal Cord Injury; Tetraplegia; Pulmonary Function; Bronchodilator
MeSH Terms: conditions — Spinal Cord Injuries; Quadriplegia | interventions — Tiotropium Bromide; Salmeterol Xinafoate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Anticholinergic Agent (Active Comparator)
  Interventions: Drug: Tiotropium
- Long Acting Beta 2 Agonist (Active Comparator)
  Interventions: Drug: Salmeterol

INTERVENTIONS:
Drug: Tiotropium — 18mcg/ capsule inhaled once daily for two weeks.
  Arms: Anticholinergic Agent
Drug: Salmeterol — 50mcg inhalation twice daily for two weeks
  Arms: Long Acting Beta 2 Agonist

SUMMARY:
To determine the acute and chronic effects of a short course of treatment on spinal cord injured (SCI) individuals with either an anticholinergic agent (tiotropium) or with a β₂ agonist (Salmeterol) on:

* Fraction of expired NO (FeNO)
* Selected Biomarkers of inflammation in exhaled breath condensates (EBC)
* Pulmonary function, as measured by pulmonary function tests and body plethysmography

ELIGIBILITY:
Inclusion Criteria:

1. Chronic Spinal Cord Injury (>1 year post-injury)
2. All American Spinal Injury Association (ASIA) classifications
3. Stable tetraplegia (level of injury C3-C8, non-ventilator dependent)
4. Age 18-65 years

Exclusion Criteria:

1. Smoking, active or history of smoking within last 6 months;
2. Active respiratory disease;
3. Known history of asthma during lifetime or recent (within 3 months) respiratory infections;
4. Use of medications known to affect the respiratory system;
5. Use of medications known to alter airway caliber;
6. Coronary heart and/or artery disease;
7. Hypertension;
8. Adrenal insufficiency;
9. Pregnancy;
10. Severe Milk Protein Allergy;
11. Lack of mental capacity to give informed consent;
12. Previous allergic reaction or hypersensitivity to salmeterol or tiotropium;
13. Individuals taking medication(s) with known /potential drug interactions or suggested therapy modification for concomitant use with salmeterol or tiotropium such as:

(1) selective alpha-/beta- blockers: carvedilol, labetalol; (2) non-selective beta-blockers: Carteolol; Levobunolol; Metipranolol; Nadolol; Penbutolol; Pindolol; Propranolol; Sotalol; Timolol); (3) CYP3A4 Inhibitors: (e.g, Atazanavir; Clarithromycin; Conivaptan; Darunavir; Delavirdine; Fosamprenavir; Imatinib; Indinavir; Isoniazid; Itraconazole; Ketoconazole; Lopinavir; Nefazodone; Nelfinavir; NiCARdipine; Posaconazole; QuiNIDine; Ritonavir; Saquinavir; Telithromycin; Voriconazole; (4) Iobenguane I 123 / Sympathomimetics: Albuterol; Aminophylline; Arformoterol; Armodafinil; Benzphetamine; Caffeine; Dexmethylphenidate; Dextroamphetamine; Diethylpropion; Dipivefrin; DOBUTamine; DOPamine; Doxapram; Dyphylline; EPHEDrine; EPINEPHrine; Fenoterol; Formoterol; Isometheptene; Levalbuterol; Levonordefrin; Lisdexamfetamine; Metaproterenol; Methamphetamine; Methylphenidate; Midodrine; Modafinil; Naphazoline; Norepinephrine; Oxymetazoline; Phendimetrazine; Phentermine; Phenylephrine; Pirbuterol; Propylhexedrine; Pseudoephedrine; Sibutramine; Terbutaline; Theophylline; Xylometazoline.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2011-08; Primary Completion 2016-03 (Estimated); Study Completion 2016-08 (Estimated)

PRIMARY OUTCOMES:
The effect of an anticholinergic agent or beta 2 agonist on the fraction of expired NO (FeNO) | Approximately 8 weeks
  This will be a crossover trial. Baseline measurements will be taken, followed by two weeks of drug intervention (Salmeterol or Tiotropium Bromide). After two weeks the subject will return for post drug measurements. There will be a wash out period of four weeks, and then the subject will return again for the baseline measurements of drug 2, followed by two weeks of intervention and a final assessment.

SECONDARY OUTCOMES:
Selected Biomarkers of inflammation(TNF-alpha,Isoprostane 8, Leukotriene B4) in exhaled breath condensates (EBC)after intervention | Approx. 8 weeks
  The subject will be randomized to receive either anticholinergic agent or long acting Beta2 agonist. Measurements of EBC will take place at baseline, 1 hr post drug administration, and two weeks after intervention. Biomarkers of inflammation will be assessed by collected exhaled breath condensates, which will subsequently be sent for biochemical analysis. Markers include Isoprostane-8, TNF-Alpha, and Leukotriene B4.
Pulmonary function, as measured by pulmonary function tests and body plethysmography | Approx. 8 weeks
  This will be a crossover trial. Baseline measurements will be taken, followed by two weeks of drug intervention (Salmeterol or Tiotropium Bromide). After two weeks the subject will return for post drug measurements. There will be a wash out period of four weeks, and then the subject will return again for the baseline measurements of drug 2, followed by two weeks of intervention and a final assessment. Pulmonary assessments include: Spirometry and Plethysmography.

CONTACTS AND LOCATIONS:
Overall Officials: Miroslav Radulovic, MD, Principal Investigator — James J. Peters VA Medical Center
Locations (2):
- United States (2):
  - Kessler Institute for Rehabilitation, West Orange, New Jersey
  - James J. Peters VA Medical Center, The Bronx, New York